CLINICAL TRIAL: NCT06144411
Title: Recording and Evaluating Preoperative Malnutrition in Electively Scheduled Adult Surgical Patients With the GLIM Criteria (GLIM-study)
Acronym: GLIM
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, B Preckel, Prof dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2023.0890
Record Dates: First submitted 2023-11-17; First posted 2023-11-22 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: prevalence of preoperative malnutrition — prevalence of preoperative malnutrition

SUMMARY:
Data about the prevalence of preoperative malnutrition according to all the five GLIM criteria among the broad range of surgical patients are lacking. The current study will investigate the prevalence of malnutrition according to all of the five GLIM criteria in electively planned surgical patients in a large academic hospital, the Amsterdam University Medical Centres, location AMC, where over 11.000 patients are operated on yearly.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective surgery at the operating theatres of the AUMC, location AMC
* Patients ≥ 18 years
* Dutch speaking
* Willing and able to sign consent for re-use of care data
* The study can be combined with other studies

Exclusion Criteria:

* Patients < 18 years
* Not speaking Dutch
* Patients who do not sign consent for re-use of care data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of electively scheduled adult surgical patients at the Amsterdam UMC, location AMC.
Sampling Method: Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
prevalence of preoperative malnutrition | preoperative
  To study the prevalence of preoperative malnutrition according to the GLIM criteria in electively scheduled adult surgical patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Hermanides, prof. dr., Principal Investigator — j.hermanides@amsterdamumc.nl
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided